CLINICAL TRIAL: NCT02747576
Title: Social Cognition and Brain Integrity in Survivors of Pediatric Medulloblastoma
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: St. Baldrick's Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: FACES
Record Dates: First submitted 2016-04-13; First posted 2016-04-22 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Medulloblastoma
Keywords: Childhood Cancer Survivor; Social-cognition; Healthy Volunteers
MeSH Terms: conditions — Medulloblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medulloblastoma Group: Medulloblastoma survivors, 30 between the ages of 12-20 years and 30 between 21-30 years.
- Control Group: Health comparison group frequency matched on age (30 between the ages of 12-20 years and 30 between 21-30 years), gender and race.

SUMMARY:
Survivors of pediatric medulloblastoma (MB) are at-risk for neurocognitive and social deficits, including specific skills such as facial affect recognition which is the ability to recognize the emotional expressions of another person. Because the underlying mechanisms of these deficits are poorly understood, the investigators propose to examine social-cognitive skills (i.e. facial affect recognition) and indices of brain integrity, including an established core neural network of face perception in MB survivors and healthy controls. By comparing these outcomes between survivors of MB and healthy controls, investigators seek to identify the areas of the brain that help individuals recognize emotions.

Primary Objective:

* To evaluate social cognition in adolescent and young adult survivors of pediatric medulloblastoma.

Secondary Objective:

* To examine indices of brain integrity and function and their association with facial affect recognition in survivors of pediatric medulloblastoma.

DETAILED DESCRIPTION:
Comprehensive social-cognitive and behavioral data will be collected and structural and functional brain imaging will be completed in an attempt to determine if disruptions to brain integrity and function caused by prior treatment of medulloblastoma directly influence social-cognition and behavior in survivors. These outcomes will be compared between survivors and age-, gender-, and race-matched healthy community controls.

Participants who meet eligibility criteria and consent will undergo neurocognitive (intelligence, attention, memory, processing speed, motor, executive function, and visuospatial) and social cognitive evaluations (affect recognition, prosody, social memory, withdrawal/isolation, loneliness, social anxiety, visuospatial, and executive function). Functional magnetic resonance imaging (fMRI) will be completed during affect identification tasks to assess activation of the core face perception network. Magnetic resonance with diffusion tensor imaging (DTI) will be obtained to quantify water diffusion within white matter tracts to assess white matter integrity and its association with functional outcomes.

ELIGIBILITY:
Inclusion Criteria - Medulloblastoma Survivors:

* Enrolled on the SJLIFE protocol at St. Jude Children's Research Hospital (SJCRH).
* Completed treatment for medulloblastoma at SJCRH.
* Infratentorial tumor location.
* Treated with craniospinal irradiation.
* ≥ 5 years post diagnosis.
* Between 12 and 30 years of age at time of enrollment.
* English speaking.

Inclusion Criteria - Controls:

* Enrolled on the SJLIFE protocol as a community control.
* Between 12 and 30 years of age at time of enrollment.
* English speaking.

Exclusion Criteria - Medulloblastoma Survivors:

* Diagnosis of a genetic disorder/pre-existing neurodevelopmental condition associated with neurocognitive or social impairment (e.g., down syndrome, autism).
* History of head injury associated with neurocognitive impairment.
* Diagnosis of a serious psychiatric condition associated with neurocognitive or social morbidities (e.g. schizophrenia).
* Currently pregnant (due to MRI studies).
* Implanted metal unsafe for MRI or medical device (i.e. pacemaker)
* Requires sedation to complete MRI.
* Legally blind or unaidable hearing loss.
* Treated for medulloblastoma <3 years of age
* Received re-irradiation to the brain.
* Completed SJLIFE HPP-19 (pilot study) at SJCRH.

Exclusion Criteria - Controls:

* No history of childhood cancer or cancer related therapy.
* First degree relative or direct friend of medulloblastoma participant.
* Diagnosis of a genetic disorder/neurodevelopmental condition associated with neurocognitive or social impairment (e.g., down syndrome, autism).
* History of head injury associated with neurocognitive impairment.
* Diagnosis of a serious psychiatric condition associated with neurocognitive or social morbidities (e.g. schizophrenia).
* Currently pregnant (due to MRI studies).
* Implanted metal unsafe for MRI or medical device (i.e. pacemaker).
* Requires sedation to complete MRI.
* Legally blind or unaidable hearing loss.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Medulloblastoma survivors enrolled in the St Jude Lifetime Cohort parent protocol will be recruited to complete comprehensive social-cognitive and neurocognitive evaluations as well as structural and functional brain imaging. Investigators will also recruit a comparison sample of healthy individuals matched on age, sex and race.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Performance on standardized measures of facial affect recognition (NEPSY-II; Advanced Clinical Solutions Social Cognition) | Within two months of participant enrollment
  Mean scores on measures of facial affect recognition will be compared between survivors of medulloblastoma and age, sex, and race matched community controls.

SECONDARY OUTCOMES:
Performance on tests of visual spatial processing and executive functioning using standardized neurocognitive assessment measures | Within two months of participant enrollment
  Means scores on measures of visual spatial processing and executive function will be compared between survivors of medulloblastoma and age, sex, and race matched community controls.
Activation of the core face perception network (lateral fusiform gyrus, inferior occipital gyri, superior temporal sulcus) using fMRI analysis | Within six months of participant enrollment
  Patterns of brain activation (i.e. hemodynamic responses) will be compared between survivors of medulloblastoma and age, sex, and race matched community controls.
White matter integrity between the nodes of the core face perception network (lateral fusiform gyrus, inferior occipital gyri, superior temporal sulcus) using DTI analysis | Within six months of participant enrollment
  Indices of white matter integrity (e.g., radial diffusivity, axial diffusivity) will be compared between survivors of medulloblastoma and age, sex, and race matched community controls.

CONTACTS AND LOCATIONS:
Overall Officials: Tara M. Brinkman, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols